CLINICAL TRIAL: NCT00163202
Title: A Multicenter, Randomized Double-Blind Study Comparing The Pleiotropic Effects Of Atorvastatin 10 Mg And 80 Mg Over A 26-Week Period In Subjects With Coronary Atherosclerosis
Brief Title: Comparative Atorvastatin Pleiotropic Effects
Acronym: CAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Collaborators: MDS Pharma Services (Industry); Bio-Inova Life Sciences International (Other)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2581065
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Coronary Arteriosclerosis; Hypercholesterolemia
MeSH Terms: conditions — Coronary Artery Disease; Hypercholesterolemia | interventions — Blood Specimen Collection; Atorvastatin

INTERVENTIONS:
Procedure: Blood samples
Drug: Atorvastatin

SUMMARY:
The primary objective of the study is to evaluate the efficacy of atorvastatin 80 mg daily as compared to atorvastatin 10 mg daily in reducing C-reactive protein levels over a 26-week treatment period in subjects with documented coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of age of majority to < 80 years
* Subjects with LDL-C > 0.5 g/L (1.29 mmol/L) and < 1.5 g/L (3.87 mmol/L), TG < 4.00 g/L (4.56 mmol/L) and hs-CRP >1.5 mg/L and < 15 mg/L
* Subjects with a documented coronary artery disease.

Exclusion Criteria:

* Female subjects of childbearing potential without contraception
* Subjects with secondary hyperlipidemia
* Diabetic subjects receiving insulin
* Subjects with a contra-indication to statin therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330
Dates: Start 2002-06; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Percentages changes of the hs-CRP between baseline (means between week-2 to -1 and week 0 (V2) values) and week 26 (V5).

SECONDARY OUTCOMES:
1/ the percentage change at visit 3 (5-week treatment), visit 4 (13-week-treatment) and visit 5 (26-week treatment) from baseline value in triglycerides, total cholesterol; HDL-cholesterol, LDL-cholesterol, apolipoprotein B 2/ the percentage change at

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (61):
- Canada (16):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Oshawa, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Weston, Ontario
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, Ste-foy, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Czechia (3):
  - Pfizer Investigational Site, Brno-Bohunice
  - Pfizer Investigational Site, Jindřichův Hradec
  - Pfizer Investigational Site, Prague
- France (31):
  - Pfizer Investigational Site, Clermont-Ferrand, Cedex
  - Pfizer Investigational Site, Langres, Cedex
  - Pfizer Investigational Site, Besançon
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Chambéry
  - Pfizer Investigational Site, Clamart
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Creil
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Évecquemont
  - Pfizer Investigational Site, Gap
  - Pfizer Investigational Site, Hénin-Beaumont
  - Pfizer Investigational Site, Le Kremlin-Bicêtre
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Metz
  - Pfizer Investigational Site, Monaco
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Mulhouse
  - Pfizer Investigational Site, Nancy
  - Pfizer Investigational Site, Nantes Saint Herblain
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Pessac
  - Pfizer Investigational Site, Poissy
  - Pfizer Investigational Site, Pontoise
  - Pfizer Investigational Site, Roubaix
  - Pfizer Investigational Site, Saint-Michel
  - Pfizer Investigational Site, Thionville
  - Pfizer Investigational Site, Toulouse
  - Pfizer Investigational Site, Tourcoing
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy
- Poland (6):
  - Pfizer Investigational Site, Bełchatów
  - Pfizer Investigational Site, Gdynia
  - Pfizer Investigational Site, Rawa Mazowiecka
  - Pfizer Investigational Site, Torun
  - Pfizer Investigational Site, Wroclaw
  - Pfizer Investigational Site, Zamość
- Romania (2):
  - Pfizer Investigational Site, Bucharest, Sector 2
  - Pfizer Investigational Site, Bucharest, Sector 5
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Volgograd
- Pfizer Investigational Site, Bratislava, Slovakia

REFERENCES:
- [Derived] Bonnet J, McPherson R, Tedgui A, Simoneau D, Nozza A, Martineau P, Davignon J; CAP Investigators. Comparative effects of 10-mg versus 80-mg Atorvastatin on high-sensitivity C-reactive protein in patients with stable coronary artery disease: results of the CAP (Comparative Atorvastatin Pleiotropic effects) study. Clin Ther. 2008 Dec;30(12):2298-313. doi: 10.1016/j.clinthera.2008.12.023. PMID 19167589